CLINICAL TRIAL: NCT03979599
Title: Safety and Efficacy of Magnesium Sulphate as an Adjuvant to Levobupivacaine in Ultra-sound Guided Transversus Abdominis Plan Block in Pediatric Abdominal Cancer Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Ahmed Kamal Sayed, Principal Investigator, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ahmed-SECI-86
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Pain
Keywords: TAP, magnisum sulphate
MeSH Terms: conditions — Pain, Postoperative | interventions — Levobupivacaine

STUDY DESIGN:
Intervention Model Description: Group A (control group): patients will receive levobupivacaine 0.25% . Group B (magnesium sulphate group): patients will receive levobupivacaine 0.25% + MgSo4 .
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: all participant will be blinded to the study drugs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- magnesium sulphate& levobupivacaine (Active Comparator): Levobupivacaine add to magnisum sulphate
  Interventions: Procedure: ultra-sound guided transversus abdominis plan block; Drug: magnesium sulphate& levobupivacaine
- levobupivacaine (Placebo Comparator): levobupivacaine
  Interventions: Procedure: ultra-sound guided transversus abdominis plan block; Drug: Levobupivacaine

INTERVENTIONS:
Procedure: ultra-sound guided transversus abdominis plan block — comparing ultrasound guided transversus abdominis plan block using combination of magnisum sulphate and levobupivacaine versus levobupivacaine
Drug: magnesium sulphate& levobupivacaine — magnesium sulphate& levobupivacaine
  Arms: magnesium sulphate& levobupivacaine
Drug: Levobupivacaine — levobupivacaine
  Arms: levobupivacaine

SUMMARY:
To study the efficacy of magnesium sulphate as adjuvant to levobupivacaine in transversus abdominis plane (TAP) block in patient undergoing abdominal cancer surgery.

DETAILED DESCRIPTION:
In this randomized study, patients with (ASA) Ӏ and ӀӀ, aged from 1 to 7 years old and their weight less than 30 Kg of both sex will undergo surgery will be enrolled.

A written informed consent from all parents are obtained

ELIGIBILITY:
Inclusion Criteria:

* patients with (ASA) Ӏ and ӀӀ physical status, aged from 1 to 7 years old and their weight less than 30 Kg of both sex will undergo surgery will be enrolled.

Exclusion Criteria:

* Children with infection, hemorrhagic disorders, hypersensitivity to the studied drugs, muscular disorders, central and peripheral neuropathy, organ dysfunction, cardiac problems and unconscious or mentally retarded patients will be excluded

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
postoperative pain management | one day
  pain will be assessed using FLACC score.The Face, Legs, Activity, Cry, Consolability (FLACC) pain score with its 0 - 10 score range will be used to assess pain immediately postoperative and then at 2, 4, 6, 8, 12, 18 and 24 hours in the postoperative period.

CONTACTS AND LOCATIONS:
Locations (1):
- south Egypt cancer institute, Asyut, Egypt